CLINICAL TRIAL: NCT00662363
Title: Lubiprostone (Amitiza®) Compared to Standard Care in the Treatment of Postoperative Opioid-induced Constipation in Inpatient Rehabilitation Patients Following Orthopedic Procedures
Brief Title: Lubiprostone (Amitiza®) Vs. Standard Care in Opioid-induced Constipation After Surgery in Inpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Christina Marciniak, Attending Physician, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00001168
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
Keywords: constipation; opioid; rehabilitation; post-operative; orthopedic
MeSH Terms: conditions — Constipation | interventions — Lubiprostone; Sennosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone and placebo Senna (Experimental): Lubiprostone (Amitiza) 24 µg po BID given with meals for 6 days with two tabs placebo Senna at noon
  Interventions: Drug: Lubiprostone
- Senna active plus Lubiprostone Placebo (Active Comparator): Senna 2 tabs daily for 6 days at noon and placebo Lubiprostone 1 Cap BID
  Interventions: Drug: Senna

INTERVENTIONS:
Drug: Lubiprostone — 24 µg po BID given with meals for 6 days
  Other Names: Amitiza
  Arms: Lubiprostone and placebo Senna
Drug: Senna — 2 tabs daily for 6 days
  Other Names: Sennasides 8.6 mg each tab
  Arms: Senna active plus Lubiprostone Placebo

SUMMARY:
Patients requiring opioids for post-operative pain control following elective orthopedic procedures which has resulted in constipation symptoms, and who are in inpatient rehabilitation will be randomized to two different treatment arms: lubiprostone or senna. Baseline scores regarding constipation and a quality of life bowel questionnaire will be compared the day following 6 days of treatment intervention.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of Lubiprostone (Amitiza) compared to standard care for the treatment of constipation in orthopedic patients receiving opioids for pain control during inpatient rehabilitation. Lubiprostone (Amitiza®) is a locally acting chloride channel activator that increases intestinal fluid, and thus increases intestinal motility. It has been approved for chronic constipation, but not in the setting of opioid-induced constipation. Senna is a stimulant laxative that increases propulsive peristaltic activity of the colon through local effects on the mucosa.

Subjects will be compared using from the Patient Assessment of Constipation (PAC) which has previously been found to be a valid and reliable way to measure constipation symptoms and clinical course. (Frank, Kleinman et al. 1999) as well as with other measures of bowel-related symptoms and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, 18 years old or greater.
2. The patient is able to provide informed consent.
3. Anticipated duration of hospitalization of at least 7 days.
4. Woman of childbearing potential must have a negative serum pregnancy test at enrollment. Exclusions for testing include two years or greater postmenopausal, hysterectomy or tubal ligation.
5. Use of opioid for post-op analgesia following orthopedic surgical procedures as defined as IV, IM, transdermal or PO opioid received within the prior 24 hours of hospitalization for pain control, and expectation that an opioid will be continued for pain control.

   * Medication may be administered on a PRN (as needed) basis or scheduled basis
   * One or greater doses has been received within the 24 hours prior to enrollment as determined by medication administration recorded from the acute care facility or RIC MAR.
6. At least one associated symptom of constipation at the time of admission, such as, but not limited to:

   * Lumpy or Hard stools
   * Feeling of incomplete evacuation of bowels
   * Abdominal cramping or pain
   * Straining with movement of bowels or painful bowel movement effort
   * Need for manual assistance to have a bowel movement

Exclusion Criteria:

1. Known allergy or sensitivity to the study medications
2. Females who are pregnant
3. Diarrhea on the day of admission
4. Diagnosis of Clostridium difficile infection during the current hospitalization
5. Pre-existing medical condition or surgical procedure, which is known to commonly lead to bowel dysfunction such as, but not limited to:

   * Crohn's disease
   * Ulcerative colitis
   * Multiple sclerosis
   * Cerebral palsy
   * Spinal Cord Injury
   * Colectomy
   * Malabsorption Syndrome
   * Irritable Bowel Syndrome
   * Abdominopelvic neoplasm (gastric, colon cancer)
   * Severe liver disease
   * Colonic or ileo-colonic resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Marciniak, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Marciniak CM, Toledo S, Lee J, Jesselson M, Bateman J, Grover B, Tierny J. Lubiprostone vs Senna in postoperative orthopedic surgery patients with opioid-induced constipation: a double-blind, active-comparator trial. World J Gastroenterol. 2014 Nov 21;20(43):16323-33. doi: 10.3748/wjg.v20.i43.16323. PMID 25473191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the inpatient population of an academic freestanding rehabilitation hospital following admission for impairments related to an orthopedic surgery.The study was approved by the local institutional review board and all subjects provided written informed consent.
Pre-assignment Details: 72 patients were recruited. There were eight who did not meet inclusion and/or exclusion criteria following consent and screening visit. Reasons for exclusion were: history of Crohn's disease (1 person), history of irritable bowel disease (1 person), diarrhea on baseline visit day (1 person), or no associated bowel symptom (5 persons).
Groups:
- Lubiprostone: Lubiprostone24 µg po BID for 6 days with placebo senna tab
- Senna: Senna 2 tabs daily for 6 days with placebo lubiprostone tabs
Period: Overall Study
Arm/Group | Lubiprostone | Senna
Started | 32 | 32
Completed | 21 (1 subject withdrew before taking any study medication) | 22 (one subject died before receiving any study med 2 subjects withdrew before taking any study med)
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Adverse Event | 0 | 3
Not completed — Discharged early from rehab | 4 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Senna | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 23 | 25 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 70.9 (11.8) | 72.2 (10.5) | 71.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Assessment of Constipation (PAC) - Symptoms (Sym)
Description: Patient Assessment of Constipation (PAC) - Change in this measure was assessed. The PAC has previously been found to be a valid and reliable way to measure constipation symptoms and clinical course. The PAC has two components. The symptom (SYM) component is composed of 12 items with score range 0-4 with lower scores indicating improvement. Scores within the two domains were separately averaged. The PAC-SYM questionnaire has shown good concurrent and clinical validity for opioid-induced constipation in a number of pain populations and has demonstrative responsiveness to treatment. There are three symptom domains within the PAC-SYM: Abdominal symptoms (4 items), rectal symptoms (3 items) and stool symptoms (5 items).
Time Frame: Baseline and Day 7, after treatment completed (6 days of treatment)
Population: All subjects randomized and who had baseline and endpoint data were included in the intention to treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Senna
Number analyzed (Participants) | 28 | 28
units on a scale | -0.22 (0.57) | -0.29 (0.58)
Statistical Analysis 1: Comparison: Lubiprostone vs Senna; Primary outcome measures chosen were between group comparisons for change on Constipation Symptom Questionnaire ratings at exit from the study. The PAC-SYM is a symptom scale where higher numbers indicate more symptoms. Change from baseline to Day 7 was calculated and larger negative differences indicated greater improvement in constipation symptoms. The PAC-QOL is a quality of life scale where higher numbers indicate better quality of life. Change from baseline to 7 days was calculated; Test type: Superiority or Other; p < 0.05, independent sample t test

2. Primary Outcome: Change in Patient Assessment of Constipation - Quality of Life
Description: The second component of the PAC is the quality of life (QOL) component.The quality of life (QOL) component consists of five items that are rated on a 0-4 scale with higher scores indicating better QOL. Scores within the domains are averaged.
Time Frame: Baseline and day 7
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lubiprostone; Senna: change in PAC-QOL
Arm/Group | Lubiprostone | Senna
Number analyzed (Participants) | 28 | 28
units on a scale | 0.99 (0.78) | .42 (0.84)

ADVERSE EVENTS:
Arm/Group | Lubiprostone | Senna
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/29
Other Adverse Events (participants affected / at risk) | 13/31 | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=31) | Senna (N=29)
patellar dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=31) | Senna (N=29)
Gastrointestinal Disorder (Gastrointestinal disorders) | 13 (22) | 8 (16)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increased INR (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Additional laxatives were frequently required for symptom control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No